CLINICAL TRIAL: NCT06301542
Title: Multimodal, Task-Aware Movement Assessment and Control Using Functional Electrical Stimulation
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, David Levine, David Levine, MD, MPH, MA- Principle Investigator, Brigham and Women's Hospital
Other Study IDs: 2020P003474
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Post-stroke
Keywords: functional electrical stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-laboratory: Patients will be brought to the laboratory for functional electrical stimulation mobility assessment.
  Interventions: Device: Functional electrical stimulation
- In-home: Patients will undergo functional electrical stimulation mobility assessment in their home.
  Interventions: Device: Functional electrical stimulation

INTERVENTIONS:
Device: Functional electrical stimulation — The FES system will be placed on the plantar flexors, dorsiflexion, and quadriceps muscles and be paired with the machine learning directed inertial measurement units.

SUMMARY:
The study aims to investigate the relationship between post-stroke adults' movement patterns and disability levels. Utilizing the functional electrical stimulation (FES) system for individualized dorsiflexor and plantar flexor assistance during gait cycles. The investigators will analyze the cycles with and without the FES system. Initially, the context-aware motion assessment and neuroprosthetic control in a clinic will transition to in-home settings as the study progresses, broadening its application for safe and effective use at home.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Capacity to consent
* Post-stroke community-dwelling adults
* Ability to follow 3-step commands

Exclusion Criteria:

* Undomiciled
* Active substance use disorder
* Active psychosis
* Domestic violence or neglect
* Inability to communicate with investigators
* Other comorbidities that prevent full participation in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty post-stroke community-dwelling adults will participate in a single in-laboratory and in-home visit, performing 5x sit-to-stand (5XSST), 5x Comfortable and 3x Fast walking speed at a 5M distance, and 5x modified Timed Up and Go (TUG). The tests will be performed twice: once with and without the task aware-neuroprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Apply functional electrical stimulation to the paretic limb of muscles of poststroke patients | 1 deployment visit in the laboratory, approximately 4 hours
  Control functional electrical stimulation applied to paretic limb muscles of patients with post-stroke hemiparesis. Based on walking-related activities, the resulting controller will stimulate the target muscle groups with properties and amplitude.

SECONDARY OUTCOMES:
Accurate motion assistance while using the functional electrical stimulation in the laboratory. | 1 deployment visit in the laboratory, approximately 4 hours
  Limb movement will be accurately detected and supplemented with functional electrical stimulation in the laboratory setting.
Accurate motion assistance while using the functional electrical stimulation in the home. | 1 deployment visit in the home, approximately 4 hours
  Limb movement will be accurately detected and supplemented with functional electrical stimulation in the home setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States